CLINICAL TRIAL: NCT06640686
Title: The Effects of Inspiratory Muscle Training on Respiratory Parameters, Trunk Control, Walking, and Functional Independence in Children With Cerebral Palsy
Brief Title: The Effects of Inspiratory Muscle Training in Children With Cerebral Palsy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Okan University (Other)
Responsible Party: Principal Investigator, Gamze Aydin, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IstanbulOkanUniv
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Cerebral Palsy
Keywords: respiratory function test; muscle strength; gait; trunk
MeSH Terms: conditions — Cerebral Palsy | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: randomized controlled study
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be blind to their group and outcomes assessor will be blind to groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inspiratory Muscle Training Group (Experimental): Inspiratory muscle training consists of strengthening exercise with threshold Inspiratory muscle training device.
  Interventions: Other: Exercise training
- Traditional Physiotherapy Group (Active Comparator): The control group will receive the traditional physical therapy program.
  Interventions: Other: Exercise training

INTERVENTIONS:
Other: Exercise training — Inspiratory muscle training for increase strength of inspiratory muscle.

SUMMARY:
Cerebral palsy (CP) is characterized by permanent or variable sensory-motor function impairments resulting from developmental anomalies or damage to the brain. Spasticity, dystonia, postural disorders, and weakened movement patterns can hinder the development of the respiratory system in children with CP. As the severity of postural disorders increases in children with CP, inadequate or improper use of respiratory muscles and insufficient ventilation reduce the mobility of the thoracic cage. The aim of study is to investigate the effects of respiratory muscle training on respiratory parameters, trunk control, walking, and functional independence in children with CP.

DETAILED DESCRIPTION:
In this prospective randomized controlled study, participants will be divided into two groups: the Inspiratory Muscle Training (IMT) group and the control group. The IMT group will receive IMT in addition to the traditional physical therapy program, while the control group will only receive the traditional physical therapy program. Respiratory muscle strength, respiratory functions, chest expansion, trunk control, walking speed and endurance, and functional independence will be assessed before and after the training.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 4 and 12 years
* Classified as levels 1, 2, and 3 according to the Gross Motor Function Classification System (GMFCS)
* Diagnosed with spastic diplegia and/or hemiplegic cerebral palsy
* Ability to cooperate during the exercises

Exclusion Criteria:

* Presence of acute or chronic respiratory diseases
* Presence of acute medical conditions
* History of active epilepsy
* Scoliosis with a Cobb angle greater than 30 degrees
* Presence of chest deformities
* Severe visual and hearing impairments

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
PP Check device | 6 months
  respiratory muscle strength will assess with device that called 'RP Check'.
spirometer | 6 months
  respiratory function test will be assess with spirometer.
trunk control mesurement scale | 6 months
  trunk control will assess with Trunk Control Measurement Scale.
10 m walking test | 6 months
  gait speed will assess with 10 meter walking test
2 minutes walking test | 6 months
  gait endurance will assess with 2 minutes walking test.
WeeFIM scale | 6 months
  functional independence will assess with WeeFIM scale.

CONTACTS AND LOCATIONS:
Overall Officials: Gamze Aydın, PhD, Principal Investigator — Okan University

IPD SHARING:
Plan to Share IPD: No